CLINICAL TRIAL: NCT06794853
Title: Mechanism of Transjugular Intrahepatic Portosystemic Shunt to Improve Sarcopenia by Down-regulation of FGF21
Brief Title: Mechanism of TIPS to Improve Sarcopenia
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiacheng Liu, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: TIPS improves sarcopenia
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia; Mechanism; Cirrhosis
Keywords: sarcopenia; cirrhosis; FGF21
MeSH Terms: conditions — Sarcopenia; Fibrosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia: Patients were diagnosed with sarcopenia on the basis of CT-quantified skeletal muscle mass index (SMI) during preoperative TIPS and postoperative follow-up. The European Association for the Study of the Liver clinical practice guidelines were used to determine the threshold value for sarcopenia, and SMI was calculated from the ratio of L3 cross-sectional area to height on CT images; those with <50 cm²/m² in men and <39 cm²/m² in women were diagnosed with sarcopenia. Patients with preoperative sarcopenia and 1-year postoperative sarcopenia who were still diagnosed with sarcopenia were in the sarcopenia group.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt
- Non-sarcopenia: Patients were diagnosed with sarcopenia on the basis of CT-quantified skeletal muscle mass index (SMI) during preoperative TIPS and postoperative follow-up. The European Association for the Study of the Liver clinical practice guidelines were used to determine the threshold value for sarcopenia, and SMI was calculated from the ratio of L3 cross-sectional area to height on CT images; those with <50 cm²/m² in men and <39 cm²/m² in women were diagnosed with sarcopenia. Patients with sarcopenia before TIPS and without sarcopenia 1 year after TIPS were considered the non-sarcopenia group.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt — All patients were treated with Transjugular Intrahepatic Portosystemic Shunt (TIPS).
  Other Names: TIPS

SUMMARY:
Sarcopenia is particularly common in patients with chronic liver disease, especially in patients with decompensated cirrhosis, where the prevalence can be more than 50%. Sarcopenia is an important risk factor for a significant increase in mortality in cirrhotic patients, and is closely associated with a high incidence of complications such as hepatic encephalopathy, ascites, and infections . Recent studies have found that TIPS not only significantly improves clinical symptoms caused by portal hypertension, but may also have a positive effect on skeletal muscle mass and function in patients. Although the effect of TIPS in improving sarcopenia has been preliminarily confirmed, its mechanism is not yet fully understood. Therefore, there is an urgent need to explore the mechanism of action of TIPS to improve sarcopenia and provide guidance for clinical treatment options.

DETAILED DESCRIPTION:
According to whether the sarcopenia improved or not in patients after TIPS, patients were divided into sarcopenia group and non-sarcopenia group, and the relationship between FGF21 levels and sarcopenia improvement in patients after TIPS was analyzed by analyzing the differences between the two groups. During the follow-up of patients after TIPS, blood samples were collected to test serum FGF21 levels and imaging examinations were performed to assess the improvement of sarcopenia; changes in nutritional status, muscle strength and function indicators were analyzed in the process of sarcopenia improvement; changes in serological indicators were analyzed in the process of sarcopenia improvement, with a focus on the serum FGF21 level; the combination of the serum FGF21 level and the muscle strength and function indicators, and evaluate their value in the prognosis of TIPS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with liver cirrhosis and needing TIPS surgical treatment;
2. Aged between 18-80 years old;
3. Able to understand and sign the informed consent form and willing to cooperate in completing the examinations and follow-up visits.

Exclusion Criteria:

1. Combination of serious cardiovascular and cerebrovascular diseases (such as acute myocardial infarction, severe heart failure, etc.);
2. Suffering from malignant tumors and in the active stage;
3. Recent (within 3 months) history of major surgeries or traumas;
4. The presence of mental illness or cognitive disorders, which are unable to cooperate with the study;
5. Undergoing other special treatments that may affect the results of the study (such as certain specific immune-suppressing agents, hormones, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cirrhosis and requiring TIPS treatment, willing to participate in this study, and meeting the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pearson Correlation between Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels and Changes in Skeletal Muscle Index (SMI) at 1 Year after Transjugular Intrahepatic Portosystemic Shunt (TIPS) | 1 year
  This endpoint evaluates whether longitudinal changes in circulating FGF21 levels after TIPS have a significant Pearson correlation with changes in skeletal muscle mass. Skeletal muscle mass is quantified by the Skeletal Muscle Index (SMI), which is measured by abdominal Computed Tomography (CT) in the unit of cm²/m² . Serum FGF21 levels are measured by Enzyme-Linked Immunosorbent Assay (ELISA) in the unit of picogram per milliliter (pg/mL). This endpoint is intended to determine the role of FGF21 in TIPS-related improvement of sarcopenia.

SECONDARY OUTCOMES:
Pearson Correlation Analysis between Changes in Handgrip Strength and Dynamic Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels after Transjugular Intrahepatic Portosystemic Shunt (TIPS) | 1 year
  This outcome measure focuses on the dynamic changes in skeletal muscle strength after TIPS, with handgrip strength as the sole assessment index, measured by an electronic handgrip dynamometer in the unit of kilogram-force (kgf). Serum FGF21 levels are measured by Enzyme-Linked Immunosorbent Assay (ELISA) in the unit of picogram per milliliter (pg/mL). Pearson correlation analysis was used to explore the linear correlation between the dynamic changes in handgrip strength and the dynamic changes in serum FGF21 levels after TIPS, so as to reflect the functional recovery status of skeletal muscle in the dimension of muscle strength.
Pearson Correlation Analysis between Changes in Gait Speed and Dynamic Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels after Transjugular Intrahepatic Portosystemic Shunt (TIPS) | 1 year
  This outcome measure focuses on the dynamic changes in physical motor function after TIPS, with gait speed as the sole assessment index, measured by the 6-meter walk test in the unit of meter per second (m/s). Serum FGF21 levels are measured by Enzyme-Linked Immunosorbent Assay (ELISA) in the unit of picogram per milliliter (pg/mL). Pearson correlation analysis was used to explore the linear correlation between the dynamic changes in gait speed and the dynamic changes in serum FGF21 levels after TIPS, so as to reflect the functional recovery status of skeletal muscle in the dimension of physical performance.
Association between Dynamic Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels and Overall Survival after Transjugular Intrahepatic Portosystemic Shunt (TIPS) | 1 year
  This endpoint investigates whether longitudinal dynamic changes in serum FGF21 levels have a significant association with the overall survival of patients after TIPS, so as to explore the prognostic value of serum FGF21 levels for the survival outcome of patients after TIPS. Cox proportional hazards regression model will be used to analyze the association between dynamic changes in serum FGF21 levels and overall survival, so as to determine whether dynamic changes in serum FGF21 levels are independent influencing factors of overall survival in patients after TIPS. Serum FGF21 levels are measured by Enzyme-Linked Immunosorbent Assay (ELISA) in the unit of picogram per milliliter (pg/mL). Overall survival is defined as the time from TIPS surgery to all-cause death or the last follow-up, assessed based on clinical follow-up records in the unit of month.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zanker J, Sim M, Anderson K, Balogun S, Brennan-Olsen SL, Dent E, Duque G, Girgis CM, Grossmann M, Hayes A, Henwood T, Hirani V, Inderjeeth C, Iuliano S, Keogh J, Lewis JR, Lynch GS, Pasco JA, Phu S, Reijnierse EM, Russell N, Vlietstra L, Visvanathan R, Walker T, Waters DL, Yu S, Maier AB, Daly RM, Scott D. Consensus guidelines for sarcopenia prevention, diagnosis and management in Australia and New Zealand. J Cachexia Sarcopenia Muscle. 2023 Feb;14(1):142-156. doi: 10.1002/jcsm.13115. Epub 2022 Nov 9. PMID 36349684